CLINICAL TRIAL: NCT00447798
Title: Project Hope: Hospital Visit is an Opportunity for Prevention and Engagement With HIV-positive Crack Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor of Sociomedical Sciences and Chair, Department of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: AAAK3156; 1R01DA017612 (NIH)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections; Crack Cocaine Use; Risky Sexual Behavior
Keywords: HIV positive; crack cocaine user; inpatient hospital setting; HIV knowledge; motivation; perceived self-efficacy; risky sexual behavior; HIV seronegativity
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevention Care Advocate (Experimental): Prevention Care Advocate (PCA) intervention contains elements based on cognitive-behavioral theories and strengths-based case management. Intervention arm participants will undergo an 8 session intervention comprised of three components: 1) An individual strengths-based case management approach aimed at motivating participants to seek or maintain their engagement with HIV primary care and drug treatment; 2) A cognitive-behavioral, skills-building approach to increase participants' risk reduction knowledge, skills, and perceived self-efficacy as well as intention to change high risk transmission behaviors; and 3) A community placement in which study participants will have the opportunity to practice their advocacy skills in prevention and care setting.
  Interventions: Behavioral: Prevention Care Advocate
- Standard of Care (No Intervention): Standard of Care (SOC) condition involves standard practice, consisting of usual inpatient/hospital services provided within normal clinical practice, plus a brief educational session consisting of the review of the topics in the "Living with HIV" brochure published by the Centers for Disease Control and Prevention (CDC).

INTERVENTIONS:
Behavioral: Prevention Care Advocate — Prevention Care Advocate: 8 Session intervention combining cognitive-behavioral skill building & strengths based case management
  Arms: Prevention Care Advocate

SUMMARY:
The proposed study uses a two-arm randomized experimental design to evaluate the efficacy of a brief, theoretically-guided, "Prevention Care Advocate" intervention with HIV-positive crack users. Study participants will be recruited from the HIV inpatient hospital wards of two inner-city hospitals that serve a similar population of HIV-positive patients: Jackson Memorial Hospital (JMH) in Miami, Florida and Grady Memorial Hospital (GMH) in Atlanta, Georgia.

DETAILED DESCRIPTION:
The proposed study uses a two-arm randomized experimental design to evaluate the efficacy of a brief, theoretically-guided, "Prevention Care Advocate" intervention with HIV-positive crack users. Study participants will be recruited from the HIV inpatient hospital wards of two inner-city hospitals that serve a similar population of HIV-positive patients: Jackson Memorial Hospital (JMH) in Miami, Florida and Grady Memorial Hospital (GMH) in Atlanta, Georgia.

This 8-session, multi-component, skills-building intervention adapted from strategies used in prior studies encourages participants to advocate prevention and receipt of primary care services for themselves and their peers. We will employ a randomized experimental design to compare the intervention's efficacy with an attention-control group.

SPECIFIC AIMS Aim 1: To evaluate the efficacy of a brief, theoretically-based intervention in reducing unprotected sexual intercourse by HIV-positive crack users recruited from the inpatient/hospital setting. The impact of the intervention on secondary outcomes including the increased use of HIV primary outpatient care and readiness for and entry to drug treatment, will also be evaluated.

Aim 2: To examine whether knowledge, motivation and perceived self-efficacy are impacted by the intervention, and if changes in these variables explain change in the behavioral outcomes of interest.

Aim 3: To determine the extent to which behavioral outcomes are maintained over time.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Sexually active
* Recruited from inpatient/hospital setting
* Crack user

Exclusion Criteria:

* HIV negative
* Not sexually active
* Not recruited from inpatient/hospital setting
* Non crack user

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2005-06; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a brief, theoretically-based intervention in reducing unprotected sexual intercourse by HIV-positive crack users recruited from the inpatient/hospital setting. | 1 year

SECONDARY OUTCOMES:
The impact of the intervention on secondary outcomes including the increased use of HIV primary outpatient care and readiness for and entry to drug treatment, will also be evaluated. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Metsch, Ph.D., Principal Investigator — University of Miami; Carlos del Rio, M.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - University of Miami Hospital & Clinics/ Jackson Memorial Hospital, Miami, Florida
  - Grady Health System-Grady Memorial Hospital, Atlanta, Georgia